CLINICAL TRIAL: NCT02830737
Title: Prospective Randomized Comparative Study on No-touch Radiofrequency Ablation Treatment of Small Hepatocellular Carcinoma
Brief Title: No-touch RFA Versus Traditional RFA for Small Hepatocellular Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, Yuelong Chai, Candidate of Doctor in Medicine, Southwest Hospital, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SWH2015LC02
Record Dates: First submitted 2016-07-05; First posted 2016-07-13 (Estimated); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Hepatocellular Carcinoma
Keywords: Small Hepatocellular Carcinoma; No-touch RFA; Traditional RFA; Recurrence rate
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Traditional RFA (Active Comparator): Using Traditional RFA for the treatment of small hepatocellular carcinoma
  Interventions: Procedure: Traditional RFA
- No-touch RFA (Experimental): Using No-touch RFA for the treatment of small hepatocellular carcinoma
  Interventions: Procedure: No-touch RFA

INTERVENTIONS:
Procedure: Traditional RFA — Radio frequency ablation via an ultrasound-guided electrode needle penetrating into the lesion center
  Other Names: RFA
  Arms: Traditional RFA
Procedure: No-touch RFA — Radio frequency ablation via an ultrasound-guided electrode needle penetrating into the tumor-free zone (within 5mm along the edge of the tumor)
  Arms: No-touch RFA

SUMMARY:
Traditional RFA treatment has been a curable therapy for small hepatocellular carcinoma (diameter≤3cm). This technique ablates the tumor via radio frequency by inserting an electrode needle directly into the tumor. This clearly violates no-touch technique based on the principle of surgical oncology. Thus the 1-year recurrence rate of the cancer is up to 30% after the treatment, and the 3-year tumor-free survival rate is only 20% - 40%. No-touch RFA treatment avoids the direct contact with the tumor that can cause the spread of cancer cells in the liver, or the Antrim spread, Therefore it has been suggested that no-touch RFA treatment reduce the recurrence rate after operation in comparison with the traditional RFA treatment. This research project aims at using the prospective randomized comparative method to compare the short-term and the long-term curative effects between no-touch RFA and traditional RFA treatments for small hepatic carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Primary hepatocellular carcinoma, according to the postoperative pathological examination as the standard, or the diagnostic criteria with reference to the 2012 American Association for the Study of Liver Diseases if the pathological evidence is not available;
2. A single tumor with a diameter ≤3cm;
3. The tumor that has not invaded the portal vein, the hepatic vein, or the secondary branch;
4. Liver function classified as Child A or B;
5. Liver reserve function test with ICG-R15 (indocyanine green retention at 15min) ≤30%, and the important organs that can function with the tolerance of RFA or partial hepatectomy;
6. No significant coagulopathy: platelet count > 50,000,000,000 /L, prolonged prothrombin time < 5 seconds;
7. Age 18 - 70 years old;
8. No acceptance of other anti-cancer therapy before the treatment.

Exclusion Criteria:

1. Complication of severe portal hypertension: a history of upper gastrointestinal bleeding, a history of severe hypersplenism, or refractory ascites;
2. Patients with extrahepatic metastasis or lymph node metastasis;
3. Patients with multiple liver tumors found from imaging exam or during the treatment;
4. Patients with pathological examinations showing the other tissue type of liver cancer after the treatment;
5. Patients who expect to receive a liver transplant;
6. Patients whose preoperative imaging exam indicates the tumor close to the gallbladder, hilar major blood vessels, bile ducts and surrounding vital organs, with a potential of serious injury by mistake or serious complications during the treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2016-01; Primary Completion 2020-08 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Recurrence Rate | 3 years

SECONDARY OUTCOMES:
Recurrence-free Survival Rate | 3 years
Overall Survival Rate | 3 years

OTHER OUTCOMES:
Number of Participants with Adverse Events | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Ma Kuansheng, Ph.D, Study Director — Institute of hepatobiliary surgery,Southwest Hospital
Locations (1):
- Institute of hepatobiliary surgery,Southwest Hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided